CLINICAL TRIAL: NCT02064894
Title: A Randomized Controlled Trial of Oral Analgesic Utilization for Pain Management of CHildhood Musculoskeletal Injuries
Brief Title: Oral Analgesic Utilization for CHildhood Musculoskeletal Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Le May, Professor and Researcher, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OUCH; MOP-125943 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-04

CONDITIONS: Musculoskeletal Injury
Keywords: children; analgesia; musculoskeletal injury; emergency; opioids
MeSH Terms: conditions — Agnosia; Emergencies | interventions — Morphine; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- oral morphine and oral ibuprofen (Experimental): Oral morphine (syrup) 0.2mg/kg (max. 15 mg) and oral ibuprofen (syrup) 10mg/kg (max. 600 mg) both administered once during the 2 hour-study time frame
  Interventions: Drug: oral morphine and oral ibuprofen
- morphine and placebo of ibuprofen (Experimental): Oral morphine 0.2mg/kg (max. 15 mg) and a placebo of ibuprofen both administered once during the 2-hour time frame of the study
  Interventions: Drug: Oral morphine
- ibuprofen and placebo of morphine (Active Comparator): Ibuprofen 10mg/kg (max. 600 mg) and placebo of morphine both administered once during the 2-hour time frame of the study
  Interventions: Drug: Oral ibuprofen

INTERVENTIONS:
Drug: oral morphine and oral ibuprofen — The combination of oral morphine and oral ibuprofen is one of the Experimental arm group
  Arms: oral morphine and oral ibuprofen
Drug: Oral morphine — Oral morphine 0.2 mg/kg (syrup) up to a maximum dosage of 15 mg, administered once during the study
  Arms: morphine and placebo of ibuprofen
Drug: Oral ibuprofen — oral ibuprofen combine to a placebo is the active comparator
  Arms: ibuprofen and placebo of morphine

SUMMARY:
Pain management for children presenting to the emergency department (ED) with an injured limb is often under-treated, even though it is known that broken arms and legs cause moderate to severe pain. Further, children are less likely to receive appropriate pain medicine than adults with similar injuries. This study aims to improve the pain treatment of children who present to the ED with a suspected fracture, or broken bone or severe sprain. The investigators will compare the use of 3 different possible medication combinations (ibuprofen alone, oral morphine alone, or combined ibuprofen and oral morphine) to determine which combination is the best at treating children's pain. The investigators also plan to verify the safety of using these different drugs to treat children's pain.

The investigators strongly believe that children's pain should be optimally treated in the ED. Adequately relieving children's pain is crucial, as inadequate pain treatment can have both short and longterm effects on the child. It also generates unnecessary stress for both the child and their caregivers/parents. Given this knowledge, the investigators feel that their study has the potential to impact care provided in EDs, and improve pain management safely, for children.

DETAILED DESCRIPTION:
Rationale. Musculoskeletal trauma (MSK-T) in children is very common and almost universally painful. Standards for children's pain management of MSK-T in the Emergency Department (ED) vary greatly between Canadian hospitals and, overall, pain is very poorly treated. This inadequate pain treatment can have significant acute and chronic negative effects. Previous studies have determined that monotherapy with ibuprofen, the most commonly prescribed oral analgesic in the ED, is likely providing inadequate pain management for children. In response to this problem, clinicians have turned back to classic oral opioids (eg morphine) and are experimenting with combination therapies. To date, few studies have focused on the efficacy of a combination of a non-steroidal anti-inflammatory drug (NSAID) (eg ibuprofen) and an opioid (eg morphine). Such a combination of analgesics is known to potentiate pain relief by blocking it at the level of both the peripheral and the central nervous system. By combining two drugs with different mechanisms of action, we may be able to provide additive analgesic effects. To our knowledge, no studies have ever studied the efficacy and safety of this combination of medication for MSK-T in pediatric EDs. Primary Hypothesis: For children with a MSK-T in the ED, the addition of morphine to ibuprofen is safe and provides better pain relief than either of the two drugs alone. Primary Research Question: For children with a MSK-T in the ED, is a combination of oral morphine (0.2 mg/kg) and oral ibuprofen (10 mg/kg) more efficacious than either of the two drugs, alone, in decreasing pain scores to <30 mm, 60 minutes after administration?

Methods. Design: This study is a double-blind, placebo-controlled, two center, three-arm, randomized clinical trial (RCT). Patients will be randomized to receive either: (a) ibuprofen (10mg/kg) + placebo or (b) morphine (0.2 mg/kg) + placebo or (c) morphine (0.2mg/kg) + ibuprofen (10mg/kg). Setting: Stollery Children's Hospital (Edmonton, AB) and CHU Ste.Justine's pediatric hospital (Montreal, PQ). Inclusion criteria: We will include children: (a) between the ages of 8 and 17 years; (b) visiting the ED with an injured upper or lower limb that is neither obviously deformed, nor neurovascularly compromised, (c) with a self-reported pain score >30 mm on a 0 to100mm Visual Analogue Scale (VAS), where 0 mm corresponds to no pain and 100 mm to the worst pain the child has experienced, and (d) who understand French or English. Sample Size: Based on previous studies, we expect that between 25-52% (Clark et al., 2007, Le May et al., 2013) of children will achieve a VAS < 30 mm at 60 minutes in the ibuprofen arm. We have conservatively set the proportion of children with VAS < 30 mm at 60 min to 50%. A sample size of 500 will be then necessary to provide at least 80% power to detect a 20% absolute difference in proportion using a two-tailed with an alpha level of 5%. In order to ensure an overall alpha level of 5%, a Bonferroni correction has been applied in order to take into account the 3 pairwise comparisons that will be performed. Primary Outcome and Measurement: The primary outcome measure will be pain intensity score under 30 mm at 60-minutes after medication administration, using the VAS). Primary Safety Outcomes: We will also assess clinical measures of safety by monitoring oxygen saturation at 30 minutes intervals, up until 120 minutes. Level of sedation/alertness, as well as the respiratory rate, of each child will be monitored at set time points in the study, up until 120 minutes. Participating children will be followed up (via phone call) at 24 hours, to record any latent side effects or adverse events. Further, acceptability of the intervention will be assessed.

Relevance: Our proposed work will be the first RCT to investigate if there is some additive effect of a bi-therapy of pain with ibuprofen and morphine. In summary, currently available research supports ibuprofen as the monotherapy agent of choice. However, given concerns regarding its ability to provide adequate relief on its own, smaller studies looked at morphine as a possible alternative combined to ibuprofen. Very few studies of analgesic combinations exist, and as such, we have yet to identify the optimal ED pain management strategy for children with MSK-T. A larger trial with careful control over principal sources of bias and a rigorous approach to safety data collection will provide clinicians with strong evidence regarding efficacy and safety on new therapeutic strategies for pain management related to MSK-T in the pediatric EDs.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 6 and 17 years
* Presenting to the ED with a musculoskeletal (MSK) trauma to either of the upper or lower limbs that is neither obviously deformed, nor neurovascularly compromised
* Self-reported pain score >29 mm on a 0 to 100mm Visual Analogue Scale (VAS)
* Able to understand French or English.

Exclusion Criteria:

* Known allergy to morphine, ibuprofen, or artificial colouring
* MSK trauma that are suspected to be due to child abuse, as determined by the triage nurse
* Inability to self-report pain
* Chronic pain issues that require daily analgesic use
* NSAID or opioid analgesic use within three hours prior to presentation to triage (Exception of acetaminophen)
* Trauma to more than one limb (except fingers and toes)
* Known hepatic or renal disease/dysfunction
* Known bleeding disorder
* Neuro-cognitive disability that precludes patients from assenting and participating to the study.
* Known history of snoring consistently for the past 5 nights

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 501 (Actual)
Dates: Start 2013-07-08 (Actual); Primary Completion 2015-06-22 (Actual); Study Completion 2015-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, PhD, Principal Investigator — St. Justine's Hospital
Locations (3):
- Canada (3):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children Hospital of Eastern Ontario, Ottawa, Ontario
  - St.Justine's Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le May S, Ali S, Plint AC, Masse B, Neto G, Auclair MC, Drendel AL, Ballard A, Khadra C, Villeneuve E, Parent S, McGrath PJ, Leclair G, Gouin S; Pediatric Emergency Research Canada (PERC). Oral Analgesics Utilization for Children With Musculoskeletal Injury (OUCH Trial): An RCT. Pediatrics. 2017 Nov;140(5):e20170186. doi: 10.1542/peds.2017-0186. Epub 2017 Oct 11. PMID 29021235

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Assessed for eligibility (n=5127) Excluded (n=4626)
  * Not meeting inclusion criteria (n=1670)
  * Excluded as per exclusion criteria (n=663)
  * Declined to participate (n=874)
  * Not evaluated (n=1144)
  * Other reasons (n=275) Randomized (n=501)
Period: Overall Study
Arm/Group | Oral Morphine and Oral Ibuprofen | Morphine and Placebo of Ibuprofen | Ibuprofen and Placebo of Morphine
Started | 99 (* Received allocated intervention (n=98) * Did not receive intervention (n=1)) | 201 (* Received allocated intervention (n=198) * Did not receive allocated intervention (n=3)) | 201 (* Received allocated intervention (n=199) * Did not receive allocated intervention (n=2))
Available at T-60 | 91 | 188 | 177
Avalaible at T-90 | 74 | 134 | 129
Completed (T-120) | 56 | 99 | 86
Not Completed | 43 | 102 | 115
Not completed — Withdrawal by Subject | 43 | 102 | 115

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Morphine and Oral Ibuprofen | Morphine and Placebo of Ibuprofen | Ibuprofen and Placebo of Morphine | Total
Number analyzed (Participants) | 91 | 188 | 177 | 456
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (2.6) | 11.7 (2.7) | 12.0 (2.7) | 11.9 (2.7)
Age, Customized [Count of Participants; unit: Participants]
  6-11 | 39 | 85 | 74 | 198
  12-17 | 52 | 103 | 103 | 258
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 82 | 84 | 204
  Male | 53 | 106 | 93 | 252
VAS score at Baseline - Continuous [Mean (Standard Deviation); unit: units on a scale] — The Visual Analogue Scale is a 0 to 100 mm continuous scale measuring the pain intensity. Score of 0="No Pain"; Score of 100="Worst imaginable pain"
  units on a scale | 60.9 (15.5) | 60.8 (15.8) | 61.0 (17.1) | 60.9 (16.2)
VAS score at Baseline stratified by pain intensity [Count of Participants; unit: Participants] — The Visual Analogue Scale is a 0 to 100 mm continuous scale measuring the pain intensity. Score of 0="No Pain"; Score of 100="Worst imaginable pain"
  Participants
    30-69 mm | 64 | 128 | 121 | 313
    > 69 mm | 27 | 60 | 56 | 143
Injury type - n(%) [Count of Participants; unit: Participants]
  Fracture | 43 | 67 | 65 | 175
  Soft tissue injury | 48 | 117 | 112 | 277
  Missing | 0 | 4 | 0 | 4
Injury location - n(%) [Count of Participants; unit: Participants]
  Wrist | 24 | 28 | 25 | 77
  Ankle | 21 | 38 | 37 | 96
  Knee | 15 | 25 | 27 | 67
  Foot | 6 | 21 | 12 | 39
  Elbow | 6 | 14 | 10 | 30
  Forearm | 6 | 11 | 12 | 29
  Other | 13 | 51 | 54 | 118

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity - Percentage of Children Who Achieved VAS < 30 mm
Description: Percentage of participants which pain intensity has decreased under 30 mm on the VAS at 60 minutes.
  The Visual Analogue Scale is a 0 to 100 mm continuous scale measuring the pain intensity. Score of 0="No Pain"; Score of 100="Worst imaginable pain"
Time Frame: 60 minutes post-analgesia
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oral Morphine and Oral Ibuprofen | Morphine and Placebo of Ibuprofen | Ibuprofen and Placebo of Morphine
Number analyzed (Participants) | 91 | 188 | 177
Percentage of participants | 33.0 [24.2 to 43.1] | 29.3 [23.2 to 36.1] | 29.9 [23.7 to 37.1]
Statistical Analysis 1: Comparison: Oral Morphine and Oral Ibuprofen vs Morphine and Placebo of Ibuprofen vs Ibuprofen and Placebo of Morphine; Test type: Superiority or Other; p = 0.81, Cochran-Mantel-Haenszel

2. Secondary Outcome: Serious Adverse Event - Side Effects and Serious Adverse Events
Description: To verify the occurence of any serious adverse event, such as respiratory depression or deep sedation, during all the time-periods of the study
Time Frame: 60, 90 and 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Morphine and Oral Ibuprofen | Morphine and Placebo of Ibuprofen | Ibuprofen and Placebo of Morphine
Number analyzed (Participants) | 91 | 188 | 177
Participants
  Side effects | 6 | 39 | 38
  Serious adverse event | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Oral Morphine and Oral Ibuprofen | Morphine and Placebo of Ibuprofen | Ibuprofen and Placebo of Morphine
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/188 | 0/177
Other Adverse Events (participants affected / at risk) | 6/91 | 39/188 | 38/177
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Morphine and Oral Ibuprofen (N=91) | Morphine and Placebo of Ibuprofen (N=188) | Ibuprofen and Placebo of Morphine (N=177)
Nausea (Gastrointestinal disorders) | 0 | 11 | 7
Abdominal pain (Gastrointestinal disorders) | 0 | 7 | 7
Drowsiness (Nervous system disorders) | 0 | 5 | 4
Fatigue (General disorders) | 2 | 4 | 4
Headache (Nervous system disorders) | 2 | 4 | 4
Others (General disorders) | 2 | 8 | 12

LIMITATIONS AND CAVEATS:
High attrition rate between the time of randomization and the 120 minutes following analgesic administration; The dose of oral morphine was within the recommended range, but higher doses have been used in other trials for MSK pain relief in children.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No